CLINICAL TRIAL: NCT00433797
Title: Prostate Phytochemical & PUFA Intervention - a Phase I/II Study
Brief Title: Dietary Intervention With Phytochemicals and Polyunsaturated Fatty Acids in Prostate Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Norwegian Cancer Society (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Rune Blomhoff, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFPI; S-06187 (REK Sør) (Other: REK Sør); 2006-18 (RRHF) (Other: Oslo University Hospital)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; PSA; antioxidant; phytochemical; tomatoes; PUFA; selenium; soy; pomegranate; grapes
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Phytochemicals; Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Tomato
  Interventions: Dietary Supplement: Prostate cancer, phytochemical and PUFA
- 2 (Experimental): Multi-diet
  Interventions: Dietary Supplement: Prostate cancer, phytochemical and PUFA
- 3 (Active Comparator): Control
  Interventions: Dietary Supplement: Prostate cancer, phytochemical and PUFA

INTERVENTIONS:
Dietary Supplement: Prostate cancer, phytochemical and PUFA — Patients with localized prostate cancer are supplemented with either tomato or a multi-diet cinsisting of grape juice, pomegranate juice, tomato, green tea, black tea, soy, selenium and PUFAs for 3 weeks.
  Other Names: PFPI

SUMMARY:
We will study the effect of dietary intervention in patients with prostate cancer. Outcomes include serum PSA kinetics, as well as biomarkers of inflammation, antioxidant status, oxidative stress and oxidative damage in blood cells, plasma, urine and prostate tissues

DETAILED DESCRIPTION:
A total of 102 patients with localized prostate cancer will be included in the study. A the time of inclusion, the participants will be randomized to three groups.

The intervention groups includes; control group, tomato group and multi-diet group. The intervention period is three week and will be completed before prostatectomy or radiation therapy.

Biomarkers og inflammation includes: acute phase proteins, cytokines, chemokines and other inflammatory mediators. Biomarker of antioxidant status includes vitamin C, vitamin E, glutathione, carotenoids, total antioxidant capacity and total phenolics. Oxidative stress markers includes; malondialdehyde, isoprostanes, 8-hydroxy-deoxyguanosine, oxidized vitamin C, total lipidperoxides (d-ROM) and protein carbonyls.

ELIGIBILITY:
Inclusion Criteria:

* Adenoarcinoma (as confirmed by histology)
* pN0/NXM0 (TNM/UICC 2002) and at least one negative prognosis factor for HDR-BT or low risk profile with the use of radical prostatectomy.
* Serum PSA< 20 ng/mL, and Gleason score =>6 or T1c- T3a, prostate volume < 60mL
* Performance status 0-1
* Normal WBC and thromocytes, Hb >11g/dl

Exclusion Criteria:

* No previous endocrine treatment
* Life expectancy > 5 år
* No possible co-morbidity (CVD, COPD, diabetes type I, vasculatory syndromes or inflammatory diseases that may affect quality of life and radiation therapy)
* Urinary retention, incontinens or IPPS score <12

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-06; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
serum prostate specific antigen | Baseline, after intervention, follow-up

SECONDARY OUTCOMES:
oxidative stress biomarkers in blood, tissue and urine | Baseline, after intervention, follow-up
antioxidant status biomarkers in blood, tissue and urine | Baseline, after intervention, follow-up
oxidative damage biomarkers in blood, tissue and urine | Baseline, after intervention, follow-up
inflammation biomarkers in blood, tissue and urine | Baseline, after intervention, follow-up
Apoptose markers in prostate tissue | Baseline, after intervention, follow-up
DNA microarrays in blood cells and prostate tissue | Baseline, after intervention, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Lilleby, MD, Principal Investigator — Rikshospitalet-Radiumhospitalet, Oslo; Sigbjørn Smeland, MD, PhD., Principal Investigator — Rikshospitalet-Radiumhospitalet, Oslo
Locations (1):
- Oslo Universuty Hospital, Radiumhospitalet and Aker, Oslo, Norway

REFERENCES:
- [Derived] Paur I, Lilleby W, Bohn SK, Hulander E, Klein W, Vlatkovic L, Axcrona K, Bolstad N, Bjoro T, Laake P, Tasken KA, Svindland A, Eri LM, Brennhovd B, Carlsen MH, Fossa SD, Smeland SS, Karlsen AS, Blomhoff R. Tomato-based randomized controlled trial in prostate cancer patients: Effect on PSA. Clin Nutr. 2017 Jun;36(3):672-679. doi: 10.1016/j.clnu.2016.06.014. Epub 2016 Jun 30. PMID 27406859